CLINICAL TRIAL: NCT04794647
Title: The Effects of Manual Therapy Applied to the Cervical Region on Balance and Proprioception in Patients With Nonspesific Neck Pain: A Randomised Placebo Controlled Study
Brief Title: The Effects of Manual Therapy on Balance and Cervical Proprioception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Zafer Günendi, Prof., Gazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24074710-604.01.01
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Neck Pain
Keywords: Mobilization, Balance, Pain, Mobility, Joint position sense.
MeSH Terms: conditions — Neck Pain; Pain | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: randomized, controlled and double blind clinical trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cervical mobilization (Experimental): 'Rotation mobilization' was applied to the symptomatic segment / segments after the detailed evaluation (symptom localization tests, cervical region safety tests, joint play tests, pain provocation/alleviation tests) in accordance with the Kaltenborn-Evjenth system in cervical region. Five series of 45-s mobilizations were performed with 15 s of rest. Each patient received 6 treatment sessions over a period of 3 week.
  Interventions: Other: Cervical mobilization
- placebo mobilization (Placebo Comparator): Placebo mobilization was applied to the cervical region in the same position and the same grip with the mobilization group. The physiotherapist put her hand on a randomly selected faset without any pushing or pulling, The duration of placebo mobilization was the same as the duration of the other group. Each patient received 6 treatment sessions over a period of 3 week.
  Interventions: Other: Placebo mobilization

INTERVENTIONS:
Other: Cervical mobilization — A kind of manual therapy tecnique applied to the cervical region
  Other Names: Manual therapy
  Arms: cervical mobilization
Other: Placebo mobilization — It was applied to the randomly selected cervical faset without any pushing or pulling in the same position and the same grip with cervical mobilization.
  Arms: placebo mobilization

SUMMARY:
Introduction: Neck pain causes disturbances in both proprioception and balance. The aim of the present study is to determine the effect of mobilization applied to the cervical region on static/dynamic balance and cervical proprioception in patients with nonspecific neck pain (NSNP).

Materials and Methods: ... patients were randomly allovated into two groups. Both grups received conventional physiotherapy program (hot pack with transcutaneous electrical nerve stimulation); additionally, the experimental group received mobilization, and the control group received placebo mobilization twice a week for 3 weeks. Before and 3 weeks later, static/dynamic balance, cervical proprioception, cervical mobility and pain were evaluated respectively with Kinesthetic Skill Training System 3000 device, joint position error test, Cervical Joint Range of Motion Device, Visual Analogue Scale.

DETAILED DESCRIPTION:
Nonspecific neck pain (NSNP) is one of the most common causes of neck pain and it occurs as a result of postural or mechanical causes without a specific musculoskeletal pathology or injury history. Neck pain leads to a decrease in the activity of the deep cervical muscle which contains a large amount of muscle spindles, with an increase in the activity of the superficial cervical muscle. Depending on the pain, chemical changes occur in the cervical receptors and differentiation in sensitivity of the muscle spindle is observed. These changes in the structures of the cervical region predispose to deterioration in the sense of proprioception, which is an important component of balance. The disruption in proprioceptive abilities causes sensori-motor defects, muscle inhibition, muscle atrophy, and muscle fatigue. Changing cervical afferent information can affect proprioception as well as balance. Both the presence of neck pain and disruptions in the proprioceptive sense may reflect negatively on balance and postural control. In a study comparing patients with neck pain with asymptomatic individuals, increases in postural sway were found in patients with neck pain, and it was stated that the increased sway was associated with the dysfunction of the postural control system.

In the light of these informations, treatment approaches that can positively contribute to proprioception and balance gain importance in patients with NSNP. Although manual therapy is used both to reduce pain, and to increase cervical mobility in patients with NSNP, the number of studies investigating the effects of manual therapy on balance and proprioception is quite insufficient.

It was thought that mobilization applied to the cervical region can improve cervical proprioception and mobility, reduce pain and contribute positively to balance. The purpose of this study is to examine the effect of mobilization applications on the balance and cervical proprioception in patients with NSNP.

ELIGIBILITY:
Inclusion Criteria:

* to be diagnosed with NSNP by a physiatrist
* to be in the age range of 18-60 years
* to have pain affected by neck movements
* to have restriction of cervical region in at least the last three weeks

Exclusion Criteria:

* Neurological or orthopedic disease that may affect balance / proprioception
* presence of neurological / inflammatory symptoms
* presence of cervical instability
* to have trauma / cervical surgery / severe osteoporosis
* to use of drugs that may affect balance (antidepressants, anticonvulsants, antihistamines, sedatives, betahistine)
* to have visual / vestibular disorder
* pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2021-01-02 (Actual); Study Completion 2021-01-02 (Actual)

PRIMARY OUTCOMES:
Balance | baseline-3rd week
  Balance measured with the Kinesthetic Ability Training System 3000 (Med-Fit Systems Inc., Fallbrook, C.A., USA) for static and dynamic balance. The increase in the balance index indicates a deterioration in balance, while the decrease in the index represents an improvement in stability.
Cervical proprioception | baseline-3rd week
  Cervical joint position error test was conducted using the CROM device in transverse plane (right and left rotation). A travel eye mask was used to blindfold the patient. The examiner held the patient's head and moved slowly to the target head position, which is 50% of the maximum cervical range of motion. When patient reached actively the target position that memorized, the difference between the target position and the position obtained was recorded. Each direction of testing was performed three times and the mean error of these trials was used in the analysis.

SECONDARY OUTCOMES:
Cervical mobility | baseline-3rd week
  Active cervical range of motion was measured with the CROM device (Cervical Range of Motion-Perfomance Attainment Associates, St. Paul, MN, 55117, United States) for each direction (flexion, extension, right and left lateral flexion, right and left rotation). It is an inclinometer system that utilizes gravity and magnetic effects.
Cervical pain | baseline-3rd week
  The visual analog scale (VAS) was used to assess patient's pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Nevin Atalay Güzel, Prof., Study Chair — Gazi Univercity
Locations (3):
- Turkey (Türkiye) (3):
  - Gazi University Faculty of Medicine, Ankara
  - Gazi Univercity, Ankara
  - Gazi University, Ankara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Binder A. The diagnosis and treatment of nonspecific neck pain and whiplash. Eura Medicophys. 2007 Mar;43(1):79-89. PMID 17369782
- [Background] Falla DL, Jull GA, Hodges PW. Patients with neck pain demonstrate reduced electromyographic activity of the deep cervical flexor muscles during performance of the craniocervical flexion test. Spine (Phila Pa 1976). 2004 Oct 1;29(19):2108-14. doi: 10.1097/01.brs.0000141170.89317.0e. PMID 15454700
- [Background] Sahrmann S, Azevedo DC, Dillen LV. Diagnosis and treatment of movement system impairment syndromes. Braz J Phys Ther. 2017 Nov-Dec;21(6):391-399. doi: 10.1016/j.bjpt.2017.08.001. Epub 2017 Sep 27. PMID 29097026
- [Background] Duray M, Simsek S, Altug F, Cavlak U. Effect of proprioceptive training on balance in patients with chronic neck pain. Agri. 2018 Jul;30(3):130-137. doi: 10.5505/agri.2018.61214. PMID 30028479
- [Background] Treleaven J. Sensorimotor disturbances in neck disorders affecting postural stability, head and eye movement control. Man Ther. 2008 Feb;13(1):2-11. doi: 10.1016/j.math.2007.06.003. Epub 2007 Aug 16. PMID 17702636
- [Background] Ruhe A, Fejer R, Walker B. Altered postural sway in patients suffering from non-specific neck pain and whiplash associated disorder - A systematic review of the literature. Chiropr Man Therap. 2011 May 24;19(1):13. doi: 10.1186/2045-709X-19-13. PMID 21609469
- [Background] Voogt L, de Vries J, Meeus M, Struyf F, Meuffels D, Nijs J. Analgesic effects of manual therapy in patients with musculoskeletal pain: a systematic review. Man Ther. 2015 Apr;20(2):250-6. doi: 10.1016/j.math.2014.09.001. Epub 2014 Sep 19. PMID 25282440
- [Background] Jun P, Page I, Vette A, Kawchuk G. Potential mechanisms for lumbar spinal stiffness change following spinal manipulative therapy: a scoping review. Chiropr Man Therap. 2020 Mar 23;28(1):15. doi: 10.1186/s12998-020-00304-x. PMID 32293493
- [Background] Lee KS, Lee JH. Effect of maitland mobilization in cervical and thoracic spine and therapeutic exercise on functional impairment in individuals with chronic neck pain. J Phys Ther Sci. 2017 Mar;29(3):531-535. doi: 10.1589/jpts.29.531. Epub 2017 Mar 22. PMID 28356648
- [Background] Fisher AR, Bacon CJ, Mannion JVH. The effect of cervical spine manipulation on postural sway in patients with nonspecific neck pain. J Manipulative Physiol Ther. 2015 Jan;38(1):65-73. doi: 10.1016/j.jmpt.2014.10.014. Epub 2014 Nov 18. PMID 25467613
- [Background] Beinert K, Lutz B, Zieglgansberger W, Diers M. Seeing the site of treatment improves habitual pain but not cervical joint position sense immediately after manual therapy in chronic neck pain patients. Eur J Pain. 2019 Jan;23(1):117-123. doi: 10.1002/ejp.1290. Epub 2018 Aug 13. PMID 29999203
- [Background] Palmgren PJ, Sandstrom PJ, Lundqvist FJ, Heikkila H. Improvement after chiropractic care in cervicocephalic kinesthetic sensibility and subjective pain intensity in patients with nontraumatic chronic neck pain. J Manipulative Physiol Ther. 2006 Feb;29(2):100-6. doi: 10.1016/j.jmpt.2005.12.002. PMID 16461168
- [Background] Heikkila H, Johansson M, Wenngren BI. Effects of acupuncture, cervical manipulation and NSAID therapy on dizziness and impaired head repositioning of suspected cervical origin: a pilot study. Man Ther. 2000 Aug;5(3):151-7. doi: 10.1054/math.2000.0357. PMID 11034885
- [Background] Law EY, Chiu TT. Measurement of cervical range of motion (CROM) by electronic CROM goniometer: a test of reliability and validity. J Back Musculoskelet Rehabil. 2013;26(2):141-8. doi: 10.3233/BMR-2012-00358. PMID 23640315
- [Background] Reddy RS, Tedla JS, Dixit S, Abohashrh M. Cervical proprioception and its relationship with neck pain intensity in subjects with cervical spondylosis. BMC Musculoskelet Disord. 2019 Oct 15;20(1):447. doi: 10.1186/s12891-019-2846-z. PMID 31615495
- [Background] Mancini M, Horak FB. The relevance of clinical balance assessment tools to differentiate balance deficits. Eur J Phys Rehabil Med. 2010 Jun;46(2):239-48. PMID 20485226
- [Background] Huskisson EC, Jones J, Scott PJ. Application of visual-analogue scales to the measurement of functional capacity. Rheumatol Rehabil. 1976 Aug;15(3):185-7. doi: 10.1093/rheumatology/15.3.185. PMID 968347